CLINICAL TRIAL: NCT06489067
Title: Study of the Thyroid Function and Echostructural Morphology in Patients Affected With Rasopathies. An Italian Multicenter Study
Brief Title: Study of the Thyroid Function and Echostructural Morphology in Patients Affected With Rasopathies (ECORAS2023)
Acronym: ECORAS2023
Status: Recruiting | Type: Observational
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Maria Felicia Faienza, Associate Professor of Pediatrics, University of Bari Aldo Moro
Other Study IDs: 1386/CEL
Record Dates: First submitted 2024-06-26; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: RASopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to evaluate the prevalence of thyroid disease, particularly with autoimmune pathogenesis (isolated hyperthyrotropinemia, hyperthyroidism, hypothyroidism, thyroid nodules) and/or morphostructural abnormalities of the thyroid gland in patients with RASopathy genetically confirmed by NGS technique (analysis of the genes: BRAF, CBL, HRAS, KRAS, LZTR1, MAP2K1, MAP2K2, MRAS, NRAS, PPP1CB, PTPN11, RAF1, RIT1, RRAS2, SHOC2, SOS1, SOS2) and to compare the data obtained in our sample with those of the general population.

The secondary aim of the study is to evaluate the association between vitamin D deficiency and/or other abnormalities of bone metabolism and thyroid disease and/or morphostructural anomalies of the thyroid gland in patients with RASopathy.

DETAILED DESCRIPTION:
All patients will undergo blood sampling aimed at studying thyroid function and autoimmunity (TSH, fT3, fT4, anti-TPO, anti-TG, anti-TSH receptor antibodies) and biomarkers of bone metabolism (calcium, phosphorus, ALP isoenzyme bone, PTH, osteocalcin, vitamin D) and a systematic color Doppler ultrasound examination of the thyroid gland in order to evaluate dimensions, echostructure and echogenicity of the thyroid parenchyma, presence of nodular lesions, vascularization and laterocervical lymphadenopathy.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed RASopathy
* Age 3-25 years

Exclusion Criteria:

* Previous radiotherapy treatments, known exposure to ionizing radiation
* Iodine deficiency
* Use of iodine-based compounds or drugs that interfere with thyroid function
* Congenital hypothyroidism/hyperthyroidism
* Severe obesity with metabolic complications

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients with genetically confirmed RASopathy
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with RASopathies presenting with thyroid function and ultrasound abnormalities compared to the general population (observational study) | 6 months
  Patients will undergo blood sampling for TSH, fT3, fT4, thyroid autoimmunity and a systematic color Doppler ultrasound examination of the thyroid gland. Setting a confidence level of 95% and a margin of error of 10%, the sample size is of 96 patients. The level of statistical significance will be α=0.05. Demographic, anthropometric and clinical data will be collected according to standard criteria for each center. Continuous variables will be reported as mean and standard deviation, or median and IQR, depending on their distribution. Categorical variables will be expressed as absolute and relative frequency (%). Parametric and non-parametric statistical tests will be performed depending on the variables and their distribution. Correlation analyses will be performed between the different variables.

SECONDARY OUTCOMES:
Number of patients with RASopathies presenting with bone disease | 6 months
  Evaluate the association between vitamin D deficiency and/or bone disease and thyroid function and/or morphostructural abnormalities of the thyroid gland in patients with RASopathy. For each patient biomarkers of bone metabolism (calcium, phosphorus, vitamin D, ALP bone isoenzyme, PTH, osteocalcin) will be evaluated in order to find a possible association with thyroid abnormalities. In order to evaluate the association between the different variables (primarily, biomarkers of bone metabolism) and the outcomes measured (thyroid dysfunction or ultrasound abnormalities), binary logistic regression models will be built, adjusting for possible confounding factors.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA FELICIA FAIENZA, MD, Principal Investigator — University of Bari
Locations (1):
- University of Bari, Bari, Italy